CLINICAL TRIAL: NCT03627754
Title: A PHASE 1, OPEN LABEL, SINGLE DOSE, PARALLEL GROUP STUDY TO EVALUATE THE PLASMA PHARMACOKINETICS OF GLASDEGIB (PF-04449913) IN HEALTHY SUBJECTS WITH NORMAL HEPATIC FUNCTION AND IN SUBJECTS WITH IMPAIRED HEPATIC FUNCTION
Brief Title: A Study to Evaluate the Effect of Hepatic Impairment on the Pharmacokinetics of Glasdegib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: B1371016
Record Dates: First submitted 2018-07-31; First posted 2018-08-13 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Hepatic Impairment
Keywords: Glasdegib; PF-04449913; Pharmacokinetics; Hepatic Impairment
MeSH Terms: interventions — glasdegib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Moderate Hepatic Impairment Group (Experimental): Subjects with Child-Pugh Classification B (score 7-9)
  Interventions: Drug: Glasdegib 100 mg single oral dose
- Severe Hepatic Impairment Group (Experimental): Subjects with Child-Pugh Classification C (score 10-15)
  Interventions: Drug: Glasdegib 100 mg single oral dose
- Normal Hepatic Function Group (Experimental): Healthy subjects with normal hepatic function
  Interventions: Drug: Glasdegib 100 mg single oral dose

INTERVENTIONS:
Drug: Glasdegib 100 mg single oral dose — A single dose of 100 mg glasdegib tablet will be administered after an overnight fast, followed by serial PK collection, discharge and follow-up.

SUMMARY:
This is a Phase 1, open-label, parallel group, single dose study to investigate the effect of moderate or severe hepatic impairment on the PK of glasdegib, compared to subjects with normal hepatic function.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, parallel group, single dose study to investigate the effect of hepatic impairment on the PK of glasdegib after administration of a single oral 100 mg dose. Subjects with moderate or severe hepatic impairment will be enrolled, followed by healthy subjects with normal hepatic function who serve as matched controls.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy or hepatically impaired female subjects of non-child bearing potential and/or male subjects who, at the time of Screening, are between the ages of 18 and 75 years, inclusive.
2. Female subjects of nonchildbearing potential must meet at least 1 of the following criteria:

   1. Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; with a serum follicle-stimulating hormone (FSH) level confirming the postmenopausal state;
   2. Have undergone a documented hysterectomy and/or bilateral oophorectomy;
   3. Have medically confirmed ovarian failure. All other female subjects (including females with tubal ligations) are considered to be of childbearing potential.
3. Body mass index (BMI) of 17.5 to 40 kg/m2; and a total body weight >50 kg (110 lb).
4. Evidence of a personally signed and dated informed consent document indicating that the subject (or a legal representative) has been informed of all pertinent aspects of the study.
5. Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Additional Inclusion Criteria for Subjects With Normal Hepatic Function:

Subjects in the normal hepatic function cohort (Cohort 3) must be considered healthy and meet all of the following additional inclusion criteria to be eligible for enrollment into the study:

1. No known or suspected hepatic impairment based on liver function tests, albumin and prothrombin time, defined as the following:

   1. ALT and AST <= upper limit of normal (ULN);
   2. Total bilirubin <= 1.5 × ULN; subjects with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is not greater than 0.5 mg/dL;
   3. Alkaline phosphatase <= ULN;
   4. Albumin within the normal range (local lab ranges);
   5. Prothrombin time (PT) within the normal range (local lab ranges).
2. Subjects must fit the demographic-matching criteria, including:

   1. A total body weight that is +/- 10 kg of the population median of the pooled hepatic impairment cohorts (Cohorts 1 and 2).
   2. An age that is +/- 5 years of the population median of the pooled hepatic impairment cohorts (Cohorts 1 and 2).
3. No known or suspected hepatic impairment.
4. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure (BP) and pulse rate (PR) measurement, 12 lead ECG or clinical laboratory tests.

Additional Inclusion Criteria for Subjects with Impaired Hepatic Function:

Subjects in the hepatic impairment cohorts (Cohorts 1 and 2) must meet the following additional inclusion criteria to be eligible for enrollment into the trial:

1. Satisfy the criteria for Class B, or C of the modified Child-Pugh Classification.
2. A diagnosis of hepatic dysfunction due to hepatocellular disease (and not secondary to any acute ongoing hepatocellular process) documented by medical history, physical examination, liver biopsy, hepatic ultrasound, computerized tomography (CT) scan, or magnetic resonance imaging (MRI).
3. Known stable hepatic impairment, defined as no evidence of clinically significant change in disease status within the last 30 days, as documented by the subject's recent medical history (eg, no worsening clinical signs of hepatic impairment, or no worsening of total bilirubin or prothrombin time by more than 50%).
4. Stable drug regimen defined as not starting a new drug or changing dosage within seven days or five half-lives (whichever is longer) prior to the dosing of investigational product. History of alcohol abuse is permissible providing that the results of alcohol test are negative at Screening and on Day -1, and the subject is willing and able to abide by the lifestyle guidelines.

Exclusion Criteria:

1. Any condition possibly affecting drug absorption (eg, gastrectomy).
2. A positive urine drug test. Subjects with hepatic impairment (Cohorts 1 and 2) will be eligible to participate if their urine drug test is positive with a drug for a prescribed substance that is not expected to interfere with the PK of glasdegib.
3. Pregnant female subjects; breastfeeding female subjects; fertile male subjects who are unwilling or unable to use at least one highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 90 days after the glasdegib dose and, refrain from sperm donation for the duration of the Study and for at least 90 days after the glasdegib dose.
4. History of sensitivity to heparin or heparin-induced thrombocytopenia.
5. Blood donation of approximately 1 pint (500 mL) or more within 56 days prior to dosing.
6. Unwilling or unable to comply with the Lifestyle Requirements.
7. Subjects who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or subjects who are Pfizer employees directly involved in the conduct of the study.
8. History of known sensitivity to glasdegib.
9. Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the dose of glasdegib (whichever is longer).
10. Subjects with a history of or current positive results for human immunodeficiency virus (HIV).
11. Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Additional Exclusion Criteria for Subjects with Normal Hepatic Function:

In addition, subjects in the normal hepatic function cohort (Cohort 3) presenting with any of the following will not be included in the trial:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies deemed relevant for participation in this study, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for males (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of Screening.
3. Screening supine BP => 140 mm Hg (systolic) or => 90 mm Hg (diastolic), following at least 5 minutes of supine rest. If BP is => 140 mm Hg (systolic) or => 90 mm Hg (diastolic), the BP should be repeated two more times and the average of the three BP values should be used to determine the subject's eligibility.
4. 12-lead ECG demonstrating QTcF >450 msec or a QRS interval >120 msec at Screening. If QTcF exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated two more times and the average of the three QTcF or QRS values should be used to determine the subject's eligibility.
5. Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of lasdegib. As an exception, acetaminophen/paracetamol may be used at doses of =<1 g/day. Limited use of nonprescription medications that are not believed to affect subject safety or the overall results of the study may be permitted on a case by case basis following approval by the sponsor. Herbal supplements and hormone replacement therapy must have been discontinued at least 28 days prior to the dose of investigational product.
6. Subjects with a history of or current positive results for hepatitis B or hepatitis C, including hepatitis B surface antigen (HepBsAg), hepatitis B core antibody (HepBcAb), or hepatitis C antibody (HCVAb).

Additional Exclusion Criteria for Subjects With Impaired Hepatic Function:

In addition, subjects in the hepatic impairment cohorts (Cohorts 1 and 2) presenting with any of the following will not be included in the trial:

1. Other clinically significant disease that contraindicates study drug or that may affect the PK of glasdegib (stable, chronic, controlled disorders such as hypertension and diabetes may be acceptable).
2. Hepatic carcinoma and hepatorenal syndrome or life expectancy <1 year.
3. Undergone porta-caval shunt surgery. NOTE: Subjects with a transjugular intrahepatic portosystemic shunt (TIPS) are permitted provided that they meet the Child-Pugh Classification criteria
4. History of gastrointestinal hemorrhage either due to esophageal varices or peptic ulcers less than one month prior to study entry.
5. Any clinically significant laboratory abnormality except for those parameters influenced by hepatic impairment. Due to potential for alteration of hepatic function in renally impaired patients, subjects must have an estimated glomerular filtration rate (eGFR) corrected for their body surface area of => 75 mL/min based on the Modification of Diet in Renal Disease (MDRD) equation, with a single repeat permitted to assess eligibility, if needed.
6. Presence of clinically active stage 3 or 4 encephalopathy.
7. Severe uncontrolled ascites and/or pleural effusion.
8. Screening blood pressure => 160 mm Hg (systolic) or => 90 mm Hg (diastolic), following at least 5 minutes of supine rest. If initial BP is => 160 mm Hg (systolic) or => 90 mm Hg (diastolic), the BP should be repeated two more times and the average of the three BP values should be used to determine the subject's eligibility.
9. Screening supine 12-lead ECG demonstrating QTcF >470 msec or a QRS interval >120 msec. If initial QTcF exceeds 470 msec, or QRS exceeds 120 msec, the ECG should be repeated two more times and the average of the three QTcF or QRS values should be used to determine the subject's eligibility.
10. Use of food, drugs, or dietary supplements that may affect the PK of glasdegib within 7 days or 5 half-lives (whichever is longer) prior to the dose of glasdegib. Use of medications that are not believed to affect subject safety and are medically necessary for the treatment and maintenance of hepatic disease and other pre-existing and/or concurrent stable comorbid conditions are permitted with approval by the sponsor. Limited use of nonprescription medications that are not believed to affect subject safety or the overall results of the study may be permitted on a case by case basis with approval by the sponsor. Herbal supplements and hormone replacement therapy must have been discontinued at least 28 days prior to the dose of investigational product.
11. Concurrent use of any of the following food or drugs known to inhibit CYP3A4 (consult the sponsor if in doubt whether a food or a drug falls into any of the above categories) within 7 days or 5 half-lives (whichever is longer) prior to the dose of glasdegib, until the completion of the last PK sample collection. Use of strong or moderate CYP3A4 inhibitors includes but is not limited to: amprenavir, aprepitant, atazanavir, boceprevir, ciprofloxacin, clarithromycin, conivaptan, darunavir, delavirdine, diltiazem, erythromycin, fluconazole, fosamprenavir, imatinib, indinavir, itraconazole, ketoconazole, lopinavir, mibefradil, miconazole, nefazodone, nelfinavir, posaconazole, ritonavir, saquinavir, telaprevir, telithromycin, troleandomycin, verapamil, voriconazole, grapefruit juice or grapefruit/grapefruit-related citrus fruits (eg, Seville oranges, pomelos). The topical use of these medications (if applicable), such as 2% ketoconazole cream, is allowed. All concomitant medications must be approved by the sponsor.
12. Concurrent use of any of the following food or drugs known to induce CYP3A4 (consult the sponsor if in doubt whether a food or a drug falls into any of the above categories) within 12 days or 5 half-lives (whichever is longer) prior to the dose of investigational product, until the completion of the last PK sample collection. Strong or moderate CYP3A4 inducers includes but is not limited to: avasimibe, bosentan, carbamazepine, efavirenz, etravirine, felbamate, modafinil, nafcillin, nevirapine, phenobarbital, phenytoin, primidone, rifabutin, rifampin, rifapentin, and St. John's wort. All concomitant medication must be approved by the sponsor.
13. Subjects with congenital long QT syndrome, medical history of Torsades de Pointes or clinically significant ventricular arrhythmias.
14. Use of PPIs, including but not limited to esomeprazole, lansoprazole, omeprazole, pantoprazole, and rabeprazole, within 5 days prior to the day of glasdegib dose (Day 1).
15. Subjects will abstain from taking lactulose or other medications which could result in diarrhea or have excessive (>2) bowel movements per day within 12 hours prior to glasdegib dosing and 12 hours post dosing.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2019-04-11 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from time 0 to infinity (AUCinf) of glasdegib | Day 1 to Day 6
  PK parameter of glasdegib to be calculated from the plasma concentration-time data
Maximum observed plasma concentration (Cmax) of glasdegib | Day 1
  PK parameter of glasdegib to be calculated from the plasma concentration-time data

SECONDARY OUTCOMES:
Incidence of adverse events | Day 1 to Day 35
  Safety and tolerability of glasdegib, including monitoring of adverse events (AE) and addition of concomitant medications; an AE is any untoward medical occurrence in a study subject administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage
Incidence of clinical laboratory abnormalities | Day 1 to Day 35
  Safety and tolerability of glasdegib including blood chemistry, hematology, coagulation, and urinalysis parameters
Incidence of vital sign abnormalities | Day 1 to Day 35
  Safety and tolerability of glasdegib including monitoring of blood pressure and pulse rate
Incidence of clinical ECG abnormalities | Day 1 to Day 35
  Safety and tolerability of glasdegib including monitoring of QT interval, RR, QTc, QTS, and PR

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - Investigational Drug Services (IDS) University of Miami Hospitals and Clinics, Research Pharmacy, Miami, Florida
  - University of Miami Division of Clinical Pharmacology, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Masters JC, LaBadie RR, Salageanu J, Li J, Shaik N. Pharmacokinetics and Safety of Glasdegib in Participants With Moderate/Severe Hepatic Impairment: A Phase I, Single-Dose, Matched Case-Control Study. Clin Pharmacol Drug Dev. 2021 Jul;10(7):707-717. doi: 10.1002/cpdd.897. Epub 2020 Dec 23. PMID 33356019
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1371016&StudyName=A+Phase+1%2C+Open+Label%2C+Single+Dose%2C+Parallel+Group+Study+To+Evaluate+The+Plasma+Pharmacokinetics+Of+Glasdegib+%28pf-04449913%29+In+Healthy+Subjects+With+Normal+Hepatic+Function+And+In+Subjects+With+Impaired+Hepatic+Function